CLINICAL TRIAL: NCT00055731
Title: Phase III Randomized Study Of Adjuvant Hormonal Therapy With And Without Docetaxel And Estramustine In Patients With Advanced Prostate Cancer Or With A High Risk Of Relapse
Brief Title: Hormone Therapy With or Without Docetaxel And Estramustine in Treating Patients With Prostate Cancer That is Locally Advanced or At High Risk of Relapse
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Sanofi (Industry); AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GETUG-12 - UC-0160/0203; CDR0000270970; EU-20238
Record Dates: First submitted 2003-03-06; First posted 2003-03-07 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Prostate Cancer
Keywords: stage III prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Goserelin; Docetaxel; Estramustine; Aspirin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Experimental)
  Interventions: Drug: bicalutamide; Drug: Goserelin Acetate; Drug: docetaxel; Drug: Estramustine phosphate sodium; Drug: acetylsalicylic acid; Procedure: conventional surgery; Radiation: radiation therapy
- Without Chemotherapy (Active Comparator)
  Interventions: Drug: bicalutamide; Drug: Goserelin Acetate; Procedure: conventional surgery; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide
  Other Names: CASODEX®
Drug: Goserelin Acetate
  Other Names: ZOLADEX®
Drug: docetaxel
  Arms: Chemotherapy
Drug: Estramustine phosphate sodium
  Arms: Chemotherapy
Drug: acetylsalicylic acid
  Other Names: Aspirin
  Arms: Chemotherapy
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Androgens can stimulate the growth of prostate cancer cells. Drugs such as nilutamide, bicalutamide, flutamide, or cyproterone may stop the adrenal glands from producing androgens. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known whether hormone therapy is more effective with or without chemotherapy in treating prostate cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of hormone therapy with or without docetaxel and estramustine in treating patients who have prostate cancer that is locally advanced or at high risk of relapse.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Locally advanced disease or at high risk for relapse
* No clinically or radiologically suspected metastases
* Prior lymphadenectomy required
* Meets at least 1 of the following criteria for poor prognosis:

  * Gleason score greater than 7
  * T3 or T4 disease
  * Prostate-specific antigen greater than 20 ng/mL
  * N1 disease

PATIENT CHARACTERISTICS:

Age

* Under 80

Performance status

* ECOG 0-2

Life expectancy

* More than 10 years

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* AST and ALT no greater than 1.5 times upper limit of normal (ULN)
* Bilirubin no greater than ULN

Renal

* Creatinine less than 1.6 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular

* No uncontrolled or severe cardiovascular disease
* No prior thrombosis

Pulmonary

* No prior pulmonary embolus

Other

* No active infection
* No intolerance to aspirin
* No other prior malignancy except basal cell skin cancer
* No physical or psychological condition that would preclude study compliance

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy

Chemotherapy

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy

* No prior hormonal therapy
* No other concurrent hormonal therapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No other concurrent anticancer therapy

Ages: 0 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 413 (Actual)
Dates: Start 2002-11-14 (Actual); Primary Completion 2010-12-21 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | From randomization to disease progression or death, up to 15 years.
  The progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.
Biological response: Prostate-specific antigen (PSA) level | 3 months
  The biological response is defined as a non-detectable serum PSA level (<0.1 ng/ml)
Cancer progression as measured by ultrasound | From randomization to disease progression, up to 15 years.
  Defined as a decrease of at least 20% in prostate volume detected by ultrasound after the neo-adjuvant treatment
Clinical progression-free survival | From randomization to disease progression or death, up to 15 years.
  The clinical progression-free survival is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse (based on bone scintigraphy, pelvic scan, or MRI evaluation).
Overall survival | From randomization to death from any cause, up to 15 years.
  The overall survival is the length of time from randomization that patients enrolled in the study are still alive. The outcome is to evaluate whether SRBT improves overall survival compared to standard of care.
Acute and late toxicity during the study | Throughout study completion, up to 15 years.
  The National Cancer Institute-Common Terminology Criteria for Adverse Events version 4.0 (NCI-CTCAE v4.0) is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Quality of life questionnaire - Core 30 (QLQ-C30) | At baseline, 3 months, and 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Fizazi, MD, PhD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (38):
- France (38):
  - Centre Paul Papin, Angers
  - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Regional Francois Baclesse, Caen
  - Polyclinique du Parc, Cholet
  - Centre Hospitalier Universitaire Henri Mondor, Créteil
  - Clinique Sainte-Marguerite, Hyères
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Centre Hospital Universitaire Hop Huriez, Lille
  - Centre Hospital Regional Universitaire de Limoges, Limoges
  - Polyclinique des Quatre Pavillons, Lormont
  - Centre Leon Berard, Lyon
  - Marseille Institute of Cancer - Institut J. Paoli and I. Calmettes, Marseille
  - CHU de la Timone, Marseille
  - Hopital Notre-Dame de Bon Secours, Metz
  - Hopital Clinique Claude Bernard, Metz
  - Centre Hospitalier General de Mont de Marsan, Mont-de-Marsan
  - Hopital Lapeyronie-CHU Montpellier, Montpellier
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Catherine de Sienne, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital de la Croix St. Simon, Paris
  - Institut Curie Hopital, Paris
  - Hopital Saint Joseph, Paris
  - Hopital Tenon, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Hospitalier de Rodez, Rodez
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - CRLCC Nantes - Atlantique, Saint-Herblain
  - Hopital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Result] Fizazi K, Lesaunier F, Delva R, Gravis G, Rolland F, Priou F, Ferrero JM, Houede N, Mourey L, Theodore C, Krakowski I, Berdah JF, Baciuchka M, Laguerre B, Flechon A, Ravaud A, Cojean-Zelek I, Oudard S, Labourey JL, Lagrange JL, Chinet-Charrot P, Linassier C, Deplanque G, Beuzeboc P, Geneve J, Davin JL, Tournay E, Culine S. A phase III trial of docetaxel-estramustine in high-risk localised prostate cancer: a planned analysis of response, toxicity and quality of life in the GETUG 12 trial. Eur J Cancer. 2012 Jan;48(2):209-17. doi: 10.1016/j.ejca.2011.10.015. Epub 2011 Nov 24. PMID 22119204
- [Result] Fizazi K, Lesaunier F, Delva R, et al.: A phase III trial of docetaxel-estramustine in high-risk localized prostate cancer (GETUG 12 trial): design, tolerance, response, and quality of life (QOL). [Abstract] 2010 Genitourinary Cancers Symposium, March 5-7, 2010, San Francisco, California. A-7, 2010.
- [Result] Fizazi K, Gravis G, Culine S: The GETUG 12 trial, a phase III randomized trial of docetaxel-estramustine in high-risk localized prostate cancer: clinical design and current status. [Abstract] 2006 Prostate Cancer Symposium, February 24-26, 2006, San Francisco, CA. A-153, 2006.
- [Derived] Fizazi K, Faivre L, Lesaunier F, Delva R, Gravis G, Rolland F, Priou F, Ferrero JM, Houede N, Mourey L, Theodore C, Krakowski I, Berdah JF, Baciuchka M, Laguerre B, Flechon A, Ravaud A, Cojean-Zelek I, Oudard S, Labourey JL, Chinet-Charrot P, Legouffe E, Lagrange JL, Linassier C, Deplanque G, Beuzeboc P, Davin JL, Martin AL, Habibian M, Laplanche A, Culine S. Androgen deprivation therapy plus docetaxel and estramustine versus androgen deprivation therapy alone for high-risk localised prostate cancer (GETUG 12): a phase 3 randomised controlled trial. Lancet Oncol. 2015 Jul;16(7):787-94. doi: 10.1016/S1470-2045(15)00011-X. Epub 2015 May 28. PMID 26028518